CLINICAL TRIAL: NCT03925298
Title: Troponin- I Elevation Predicts Outcome After Thrombolysis in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, rania sanad, Principal Investigator, Zagazig University
Other Study IDs: ZU-IRB#5335\ 24-6-2018
Record Dates: First submitted 2019-04-17; First posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Cerebrovascular Accident
Keywords: acute ischemic stroke; troponin-I; outcome; intravenous thrombolytic therapy
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Serum troponin I (T-I) was collected at hospital admission at the emergency department, before any treatment. Serum samples from patients were drawn using standard venipuncture techniques. Blood samples were left to clot for 4 hours at room temperature, then centrifuged to obtain the serum which was stored frozen at (-20C). Serum T-I levels were quantified in an enzyme-linked immune-sorbent assay technology (ELISA) following manufacturer's instructions (ALPCO, 26G Keewaydin Drive, Salem NH03079, USA). Upper reference limit for apparently healthy individuals is <0.01μg/l.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: participants with elevated serum troponin level (≥0.01μg/L)
- group 2: those with normal serum troponin level (<0.01μg/L)

SUMMARY:
Elevated level of serum troponin (T-I) has been regarded as a prognostic biomarker of poor outcome in acute ischemic stroke. However, its role in outcome in thrombolysed ischemic stroke patients remains uncertain. The aim of this study was to evaluate the role of T-I as a predictive biomarker of short-term outcome in thrombolysed ischemic stroke participants.

DETAILED DESCRIPTION:
Elevated level of serum troponin (T-I) has been regarded as a prognostic biomarker of poor outcome in acute ischemic stroke. However, its role in outcome in thrombolysed ischemic stroke patients remains uncertain. The aim of this study was to evaluate the role of T-I as a predictive biomarker of short-term outcome in thrombolysed ischemic stroke patients. Methods: This study included 72 acute ischemic stroke participants were treated with intravenous thrombolytic therapy. All participants were subjected to general and neurological evaluation including assessment of stroke severity using National Institute of Health Stroke Scale (NIHSS) at admission and investigations including measurement of serum level of T-I on admission. Outcome was assessed three months after stroke onset using NIHSS and modified Rankin scale (mRS).

ELIGIBILITY:
Inclusion Criteria:

* Participants were eligible for inclusion in the study if they had evidence suggesting acute ischemic stroke that lasted for ≤ 4.5 hours .
* Those Participants were treated with intravenous thrombolytic therapy ((recombinant tissue plasminogen activator (rt-PA)).

Exclusion Criteria:

* Those who had hemorrhagic stroke
* participants presented with acute myocardial infarction, cerebrovascular stroke in the previous three months.
* serious head trauma in the previous three months.
* urinary tract, lung, or gastrointestinal hemorrhage within the three weeks.
* serious trauma or major surgery within the previous two weeks.
* lumbar or arterial puncture at a non-compressible site within one week.
* those received heparin within 48 hours, resulting in an activated partial thromboplastin time greater than the upper limit of normal.
* systolic pressure > 185 mmHg or diastolic pressure > 110 mmHg.
* blood glucose <50 or > 400 mg/dL.
* current use of anticoagulants with an International Normalized Ratio > 1.7 or prothrombin time>15 sec; platelet count < 100,000/mm3.
* pregnancy; serious heart, lung, kidney or other organ dysfunction.
* allergy to active ingredients of rt-PA; patients with > 4.5 hours from the last time known to be asymptomatic.
* those in whom troponin was not measured at admission were excluded from the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eighty one thrombolysed ischemic stroke patients were enrolled in this study. Participants who did not complete the study (9 Participants were lost during follow up) were eliminated. So the study included seventy two Participants (34 males and 38 females) who fulfilled the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
good neurological Outcome after thrombolysis | three months
  Neurological Outcome was assessed by National Institute of Health Stroke Scale (NIHSS) . good outcome (neurological improvement) was defined as 8 points improvement in NIHSS
poor neurological Outcome after thrombolysis | three months
  Neurological Outcome was assessed by the modified Rankin Scale (mRS). The modified Rankin Scale consists of 6 grades, from 0 to 5, with the best score 0 (corresponding to no symptoms) and the worst score 5 (corresponding to severe disability).
  Poor outcome was defined as death or disability (mRS scores ≥2).

IPD SHARING:
Plan to Share IPD: Yes
after publishing the manuscript in the Egyptian journal of neurology. psychiatry and neurosurgery
Supporting Information: Study Protocol, SAP
Time Frame: after publishing the manuscript in the Egyptian journal of neurology. psychiatry and neurosurgery
Access Criteria: after publishing the manuscript in the Egyptian journal of neurology. psychiatry and neurosurgery
URL: http://ejnpn.springeropen.com